CLINICAL TRIAL: NCT02143349
Title: Investigation of Appetite Suppressant Properties Associated With Coleus Forskohlii in Overweight and Obese Individuals
Brief Title: The Effect of Coleus Forskohlii Extract on the Risk Factors of Metabolic Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olive Lifesciences Pvt Ltd (Industry)
Collaborators: College of Health and Biomedicine, Victoria University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ACTRN12614000305628
Record Dates: First submitted 2014-05-17; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: obesity; herbal remedies; metabolic disorders
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coleus forskohlii extract (Experimental): Ingestion of 250 mg capsle (Coleus forskohlii extract) twice a day for 12 weeks
  Interventions: Dietary Supplement: Coleus forskohlii extract
- Placebo (Placebo Comparator): Ingestion of 250 mg capsule (placebo) twice a day for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coleus forskohlii extract — Ingestion of 250 mg Coleus forskohlii extract capsule twice a day for 12 weeks
  Arms: Coleus forskohlii extract
Other: Placebo — Ingestion of 250 mg placebo capsule twice a day for 12 weeks
  Arms: Placebo

SUMMARY:
Coleus forskohlii extract contains the bioactive compound, forskolin. Preliminary studies have shown that forskolin can increase fat metabolism thus reduce fat accumulation in both animals and humans. It has been suggested that forskolin may also suppress appetite thus reduce energy intake and results in weight loss. This study will evaluate the appetite suppressant properties of Coleus forskohlii extract. In addition the effect on central obesity and risk factors of metabolic syndrome will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Both Australian males and females, age 20-60 years, Overweight or obese (BMI >25), waist circumference of > 94 cm (male), waist circumference of >80 cm (female)

Exclusion Criteria:

* Cigarette smoker, hypertension, all types of heart, liver and kidney disease, pregnancy, lactating, Type 1 diabetes and weight loss medication.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
changes in appetite will be assessed using visual analogue scale; blood hormone levels will also be measured using commercial kits. | Baseline and 12 weeks

SECONDARY OUTCOMES:
reduction in central obesity - waist circumference will be measured on fortnight basis | 12 weeks

OTHER OUTCOMES:
alterations in blood lipids. This will be measured using commercial kits | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- College of Health and Biomedicine Victoria University, St Albans, Victoria, Australia

REFERENCES:
- [Background] obesity
- [Background] Shivaprasad HN, Gopalakrishna S, Mariyanna B, Thekkoot M, Reddy R, Tippeswamy BS. Effect of Coleus forskohlii extract on cafeteria diet-induced obesity in rats. Pharmacognosy Res. 2014 Jan;6(1):42-5. doi: 10.4103/0974-8490.122916. PMID 24497741
- See also: Coleus forskohlii extract — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0066428895&QV1=COLEUS+FORSKOHLII+EXTRACTS